CLINICAL TRIAL: NCT06418854
Title: Dengue Vaccine Hesitancy Among International Travelers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Thundon Ngamprasertchai, MD, Assoc.Prof., Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MUTM-2024-030-01
Record Dates: First submitted 2024-05-08; First posted 2024-05-17 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-01

CONDITIONS: Vaccine Hesitancy
Keywords: Dengue vaccine hesitancy; International travelers; 5C(Confidence, Complacency, Constraints, Risk calculation, Collective responsibility) model
MeSH Terms: conditions — Vaccination Hesitancy | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Non-endemic international travelers (Experimental)
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Adapted design questionnaire to estimate the vaccine hesitancy specifically for dengue vaccine

SUMMARY:
The goal of this cross-sectional study is to study dengue vaccine hesitancy among 390 international travelers who visit the Hospital for Tropical Diseases, Bangkok, and three public sites which are the area near the Grand Palace, Khaosan Road, and the snake farm at Queen Saovabha Memorial Institute. The main question it aims to answer is what are the factors associated with the dengue vaccine hesitancy among non-endemic international travelers visiting Thailand.

Participants will do the questionnaire consists of three parts

1. Questionnaire to estimate vaccine hesitancy on each 5 domains.
2. Knowledge about dengue infection and vaccination
3. Demographics data of the participants The study prioritizes ethical considerations, confidentiality, and data management to ensure participant welfare and data security.

DETAILED DESCRIPTION:
Rationale:

Dengue, a disease caused by the flavivirus and characterized by four distinct serotypes, stands as a substantial public health concern, with an estimated 390 million infections occurring worldwide annually. Clinical manifestations range from mild febrile illness to severe dengue, with secondary infections carrying a heightened risk due to antibody-dependent enhancement (ADE). The incidence of dengue among travelers to endemic areas is around one percent monthly, influenced by factors like exposure duration, seasonality, and traveler activities. Despite lacking a specific treatment, vaccination has emerged as a promising preventative measure. However, the initial vaccines licensed in the market have demonstrated limited efficacy. Vaccination in a naïve population has been associated with an increased likelihood of severe disease during the initial natural dengue infection. The recently licensed second dengue vaccine requires further information before comprehensive guidelines for usage in travelers can be established.

The rise of vaccine hesitancy, marked by reluctance or refusal, poses a growing concern, potentially leading to low vaccine coverage and emerging outbreaks. The literature about dengue vaccine hesitancy is very scarce because, unlike measles or COVID-19(CoronaVirus Disease of 2019), the efficacy of the dengue vaccine does not prove itself as a highly recommended option to prevent the disease. However, the controversial incident with the first dengue vaccine seemed to embed significant hesitation in both dengue and other vaccinations as well. Furthermore, proactive preparation for the prospective integration of the dengue vaccine into the national immunization program or its designation as a recommended vaccine for travelers is also crucial. This research aims to determine dengue vaccine hesitancy and its associated factors among non-endemic international travelers visiting Thailand, providing valuable insights for future vaccine recommendations and discussions.

Objectives:

1. To study the dengue vaccine hesitancy among non-endemic international travelers visiting Thailand.
2. To assess the factors associated with the dengue vaccine hesitancy among non-endemic international travelers visiting Thailand.

Methodology:

The cross-sectional study will recruit 390 international travelers who visit the Hospital for Tropical Diseases, Bangkok, and three public sites which are the area near the Grand Palace, Khaosan Road, and the snake farm at Queen Saovabha Memorial Institute. Data collection involves a one-time gathering of information, with eligible participants willing to provide informed consent. The questionnaire can be done both paper-based and online-based (JOTFORM), which takes time around 10-15 minutes. The questionnaire consists of 3 main parts including, a question assessing dengue vaccine hesitancy, knowledge about dengue vaccination, and demographic data. The questionnaire for estimating dengue vaccine hesitancy was derived from previous literature and validated with the pilot cohort of 20 participants. The study prioritizes ethical considerations, confidentiality, and data management to ensure participant welfare and data security.

ELIGIBILITY:
Inclusion Criteria

* Male and female international travelers from dengue-non-endemic countries
* Age ≥18 years old
* Able to read and understand English questionnaire
* Willing to participate in the study Endemic countries of dengue will be defined as all countries in the ASEAN(Association of Southeast Asian Nations) economic community countries, Central and South American countries except Chile, and ten countries in Eastern Mediterranean and Africa showing high frequency of dengue transmission according to WHO(World Health Organization) and ECDC(European Centre for Disease Prevention and Control) data(Yemen, Egypt, Sudan, Eritrea, Djibouti, Tanzania, Kenya, Ethiopia, Somalia, Burkina Faso). Non-endemic countries refer to all the other countries apart from endemic countries.

Exclusion Criteria

* Travelers who are visiting the hospital for dengue vaccination or dengue infection or dengue-like symptoms, which is defined as acute fever with one of the following; rash, myalgia, headache, nausea, vomiting, retro-orbital pain.
* Participants who are expatriate workers or lived in Thailand or other Southeast Asia countries for more than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Dengue vaccine hesitancy score | Baseline
  Spectrum of the dengue vaccine hesitancy score will be assessed by the 15 items questionaire with 7 likert scales adapting from 5C determinants of the vaccine hesitancy. The score ranging from 3-45 for each 5 domains. Higher score will represent stronger impact for each determinants; the positive determinants are confidence and collective responsibility while negative determinants are constraints, complacency, and calculation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Tropical Diseases, Bangkok, Ratchathewi, Thailand